CLINICAL TRIAL: NCT07337070
Title: Chronological Versus Non-Chronological Method in Phacoemulsification Training for Ophthalmology Residents
Brief Title: Chronological Versus Non-chronological Phacoemulsification Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Abdalsadek Ahmed Sinjab, Lecturer of Ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-25-12-9PD
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Age-related Cataract
Keywords: Phacoemulsification; Learning curve in cataract surgery; Training of ophthalmology residents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Procedure: Chronological phacoemulsification training
- Group B (Active Comparator)
  Interventions: Procedure: Non-Chronological phacoemulsification training

INTERVENTIONS:
Procedure: Chronological phacoemulsification training — Residents trained step-by-step in the natural order of phacoemulsification (incision, capsulorhexis, hydrodissection, phacoemulsification, irrigation/aspiration, IOL implantation, wound closure).
  Arms: Group A
Procedure: Non-Chronological phacoemulsification training — Residents trained initially on selected steps (e.g., wound construction, IOL implantation, cortical cleanup) before progressing to more critical steps such as capsulorhexis and phacoemulsification
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare between two methods used in training residents on phacoemulsification. The residents were classified into two groups; the first group were trained on surgical steps in a chronological order, while the second groups in non-chronological order. The outcomes included surgical competency, success rate and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 years or more with age-related cataract, and prepared for phacoemulsification.

Exclusion Criteria:

* Dense nuclear cataract grade IV or dense.
* Intumescent cataract
* Complicated and traumatic cataract
* Zonular dehiscence
* Poor pupillary dilatation
* Coexisting ocular disorder (glaucoma, PEX, uveitis,central corneal opacity….)
* Endothelial cell count 2000 or less
* Axial length 21 mm or less, 26 mm or more.
* Previous intraocular surgery
* Poor vision in the fellow eye due to irreversible condition (6/60 or less)
* Previous complicated cataract surgery in fellow eye.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Success rate | From enrollment till three months after the last surgery

SECONDARY OUTCOMES:
Incidence of complications | From enrollment till 3 months after the last surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: By April 2026 and forever
Access Criteria: Will be uploaded at clinical trail registration record or upon request via email